CLINICAL TRIAL: NCT07406542
Title: A Randomized, Open-Label, Parallel-Control, Multicenter Phase III Clinical Study of SYS6010 Versus Investigator's Choice Chemotherapy in HER2-Negative, EGFR-Positive Recurrent or Metastatic Breast Cancer
Brief Title: A Phase III Study of SYS6010 Versus Chemotherapy in HER2-Negative, EGFR-Positive Recurrent or Metastatic Breast Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Megalith Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYS6010-021
Record Dates: First submitted 2026-01-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Recurrent or Metastatic Breast Cancer
MeSH Terms: conditions — Recurrence; Breast Neoplasms | interventions — eribulin; Capecitabine; Gemcitabine; Vinorelbine

STUDY DESIGN:
Intervention Model Description: multicenter, randomized, open-label, parallel-control Phase III clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYS6010 (Experimental)
  Interventions: Drug: SYS6010
- Investigator's Choice of Chemotherapy (Active Comparator): eribulin, capecitabine, gemcitabine, or vinorelbine
  Interventions: Drug: Investigator's Choice of Chemotherapy (eribulin, capecitabine, gemcitabine, or vinorelbine)

INTERVENTIONS:
Drug: SYS6010 — SYS6010, intravenous infusion
  Arms: SYS6010
Drug: Investigator's Choice of Chemotherapy (eribulin, capecitabine, gemcitabine, or vinorelbine) — eribulin 1.4 mg/m² Intravenous infusion Administered on Day 1 and Day 8, Q3W Capecitabine 1000-1250 mg/m² orally Twice daily, Days 1-14, Q3W Gemcitabine 1000 mg/m² Intravenous infusion Administered on Days 1 and 8, Q3W Vinorelbine 25 mg/m² Intravenous infusion Administered on Day 1 and Day 8, Q3W
  Arms: Investigator's Choice of Chemotherapy

SUMMARY:
This study is a multicenter, randomized, open-label, parallel-control Phase III clinical trial enrolling patients with unresectable HER2-negative, EGFR-positive recurrent/metastatic breast cancer who have previously failed first- or second-line chemotherapy. It aims to compare the efficacy and safety of SYS6010 monotherapy versus investigator-selected chemotherapy.The study plans to enroll approximately 400 subjects, randomly assigned in a 1:1 ratio to the treatment arm and control arm(Investigator's choice of standard chemotherapy regimen, including eribulin, capecitabine, gemcitabine, or vinorelbine).

DETAILED DESCRIPTION:
This is a randomized, open-label, multicenter study designed to evaluate the efficacy and safety of SYS6010 injection versus investigator's choice of standard chemotherapy in patients with unresectable locally advanced or metastatic breast cancer that is HER2-negative with centrally confirmed EGFR expression, who have received at least one but no more than two prior lines of systemic chemotherapy for advanced or metastatic disease.

Approximately 400 patients will be enrolled and randomized in a 1:1 ratio to receive either SYS6010 injection or investigator's choice of chemotherapy. Patients randomized to the experimental arm will receive SYS6010 injection。 Patients randomized to the control arm will receive investigator's choice of standard chemotherapy, which may include eribulin, capecitabine, gemcitabine, or vinorelbine, administered per local label and institutional standard practice.

This study aims to determine whether SYS6010 provides clinically meaningful improvement in PFS compared with standard chemotherapy in patients with HER2-negative, EGFR-expressing advanced breast cancer.

The primary endpoint is progression-free survival (PFS) assessed by a blinded independent central review (BICR) per RECIST v1.1.

Secondary endpoints include overall survival (OS), investigator-assessed PFS, objective response rate (ORR), clinical benefit rate (CBR), disease control rate (DCR), duration of response (DoR), safety and tolerability, quality of life, pharmacokinetics, and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years inclusive, no gender restrictions.
2. Histopathologically confirmed breast cancer at an unresectable recurrent or metastatic stage, requiring: a) HER2-negative; b) EGFR-positive expression.
3. Subjects must have received 1 to 2 lines of systemic chemotherapy regimens during the unresectable advanced or metastatic stage.
4. At least one measurable lesion confirmed by CT or MRI according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Brain metastases are evaluated only as non-target lesions. Patients with skin lesions only are ineligible.
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
6. Expected survival ≥3 months.
7. Adequate major organ function status within 7 days prior to first study drug administration.
8. Subjects must agree to use effective contraception from informed consent signing until the protocol-specified time after last dose; females must not be lactating and males must refrain from sperm donation during this period. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to the first study drug administration. Female subjects must not be lactating.
9. Voluntarily participate in this clinical study, understand the research procedures, and be able to sign a written informed consent form.

Exclusion Criteria:

1. Presence of cancerous meningitis, spinal cord compression, or active central nervous system metastases. Active central nervous system metastases are specifically defined as untreated, symptomatic, or requiring corticosteroids/anticonvulsants to control related symptoms; except for cases stable for at least one month following treatment for brain metastases and having discontinued corticosteroids/anticonvulsants for >2 weeks.
2. Poorly controlled pleural effusion, pericardial effusion, or ascites requiring frequent drainage or medical intervention (including clinically significant recurrence requiring additional intervention within 2 weeks prior to enrollment).
3. History of other malignancies within 3 years prior to first use of study drug, except for: cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate carcinoma in situ, papillary thyroid carcinoma, and cervical carcinoma in situ
4. Prior treatment with topoisomerase I inhibitors (including ADCs)
5. Prior treatment with EGFR-targeted ADCs or monoclonal antibodies
6. Known hypersensitivity to any component of SYS6010 or to humanized monoclonal antibody products
7. Adverse events from prior antitumor therapy not recovered to ≤ Grade 1 according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 (excluding Grade 2 alopecia, asymptomatic laboratory abnormalities, etc., deemed safe by the investigator).
8. Patients with inadequate washout periods for prior medications or treatments, as specified in the protocol, prior to the first administration of the study drug. 9. History of severe cardiovascular or cerebrovascular disease.

10. Clinically significant pulmonary impairment due to pulmonary complications. 11. History of interstitial lung disease (ILD)/non-infectious pneumonia requiring glucocorticoid therapy, current ILD/non-infectious pneumonia, or inability to exclude ILD/non-infectious pneumonia based on imaging at screening.

12. Subjects with active inflammatory bowel disease, gastrointestinal obstruction, active peptic ulcer, recent (within 4 weeks) gastrointestinal bleeding, gastrointestinal perforation, or severe gastrointestinal conditions such as abdominal abscess (excluding those with a history of resolved conditions).

13. Severe infection within 4 weeks prior to first use of the investigational drug, including but not limited to: bacteremia requiring hospitalization, severe pneumonia, active tuberculosis infection, or requiring oral or intravenous antibiotic, antifungal, or antiviral therapy due to infection within 2 weeks prior to first dosing (except for prophylactic use).

14. Uncontrolled diabetes (fasting blood glucose ≥10 mmol/L and/or HbA1c ≥8%). 15. Active hepatitis B, active hepatitis C virus infection, or active syphilis infection.

16. Human immunodeficiency virus (HIV) infection diagnosed as acquired immunodeficiency syndrome (AIDS).

17.Other conditions deemed unsuitable for participation in this clinical trial by the investigator (e.g., uncontrolled psychiatric disorders or anticipated poor compliance).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
PFS | Randomization up to approximately 36 months
  PFS(progression free survival) assessed by BICR based on RECIST v1.1 criteria

SECONDARY OUTCOMES:
OS (overall survival) | Randomization up to approximately 60 months
  Overall survival is defined as the time from randomization to death from any cause.
Progression-Free Survival (PFS) Assessed by Investigator | Randomization up to approximately 36 months
  Progression-free survival assessed by the investigator is defined as the time from randomization to the first documented disease progression or death from any cause, whichever occurs first, according to RECIST version 1.1.
Objective Response Rate (ORR) | Randomization up to approximately 36 months.
  Objective response rate is defined as the proportion of patients achieving a confirmed complete response (CR) or partial response (PR) according to RECIST version 1.1, as assessed by both BICR and the investigator.
Disease Control Rate (DCR) | Randomization up to approximately 36 months.
  Disease control rate is defined as the proportion of patients achieving complete response (CR), partial response (PR), or stable disease (SD) according to RECIST version 1.1, as assessed by both BICR and the investigato.
Duration of Response (DoR) | Randomization up to approximately 36 months
  Duration of response is defined as the time from the first documented evidence of complete response (CR) or partial response (PR) until the first documented disease progression or death from any cause, whichever occurs first, according to RECIST version 1.1, as assessed by both BICR and the investigator.
Mean change from baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Randomization up to approximately 36 months
  Health-related quality of life will be assessed using the EORTC QLQ-C30 according to the Scoring Manual.
  The EORTC QLQ-C30 consists of functional scales, symptom scales, and a Global Health Status/Quality of Life scale, with scores linearly transformed to a 0 to 100 scale.
  For functional scales and the Global Health Status/Quality of Life scale, higher scores indicate better functioning or quality of life.
  For symptom scales, higher scores indicate greater symptom burden. The outcome measure is the change from baseline in the selected QLQ-C30 scale scores at post-baseline assessments.
Mean change from baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Breast Cancer Module 42 (EORTC QLQ-BR42) | Randomization up to approximately 36 months
  Breast cancer-specific quality of life will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Breast Cancer Module (EORTC QLQ-BR42), a supplementary module to the EORTC QLQ-C30, scored according to the EORTC QLQ-BR42 Scoring Manual.
  Scores for each scale are linearly transformed to a 0 to 100 scale. For functional scales, higher scores indicate better functioning; for symptom scales, higher scores indicate greater symptom burden.
  The outcome measure is the change from baseline in each BR42 scale score at post-baseline assessments.
AEs and SAEs | From first dose of study treatment until 30 days after the last dose.
  Incidence and severity of AEs and SAEs (per CTCAE 5.0), and clinically significant abnormal laboratory findings.
Maximum Observed Plasma Concentration (Cmax) of SYS6010 | Up to approximately 168 hours after the first dose of SYS6010.
  The maximum observed plasma concentration (Cmax) of SYS6010 will be determined based on measured plasma concentrations following study drug administration, using standard non-compartmental pharmacokinetic analysis methods.
Area Under the Plasma Concentration-Time Curve (AUC) of SYS6010 | From the first dose up to approximately 168 hours post-dose.
  The area under the plasma concentration-time curve (AUC) of SYS6010 will be calculated based on measured plasma concentration-time data following study drug administration, using non-compartmental pharmacokinetic analysis.
Number of Participants With Anti-Drug Antibodies (ADAs) to SYS6010 | From baseline (prior to first dose) up to approximately 30 days after the last dose of SYS6010.
  Immunogenicity will be assessed by the incidence of anti-drug antibodies (ADAs) to SYS6010. Based on blood samples collected at predefined time points during the study.